CLINICAL TRIAL: NCT06728774
Title: Cognitive Rehabilitation for Veterans With MDD-related Cognitive Functioning Deficits, w/ Joren Adams
Brief Title: Cognitive Rehabilitation for Veterans With MDD-related Cognitive Functioning Deficits
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Portland VA Medical Center (U.S. Federal Agency)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Joren Adams, Graduate Researcher, Portland VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6316
Record Dates: First submitted 2024-11-18; First posted 2024-12-11 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Major Depressive Disorder (MDD); Cognitive Dysfunction
Keywords: Veterans; Cognitive Rehabilitation; Group Intervention
MeSH Terms: conditions — Depressive Disorder, Major; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivationally Enhanced Compensatory Cognitive Training for Major Depressive Disorder (Experimental): Motivationally Enhanced Compensatory Cognitive Training for Major Depressive Disorder (ME-CCT-MDD) is a manualized group-based behavioral intervention (8 weeks, 2 hour per week) designed to improve cognitive functioning in Veterans with Major Depressive Disorder (MDD) and cognitive complaints.
  Interventions: Behavioral: Motivationally Enhanced Compensatory Cognitive Training for Major Depressive Disorder (ME-CCT-MDD)
- Goal-focused Supportive Contact (Active Comparator): Goal-focused Supportive Contact (GSC) is a group therapy intervention that provides the same frequency (8 weeks , 2 hours per week) and amount of therapist and other group member contact as ME-CCT-MDD.
  Interventions: Behavioral: Goal-focused Supportive Contact

INTERVENTIONS:
Behavioral: Motivationally Enhanced Compensatory Cognitive Training for Major Depressive Disorder (ME-CCT-MDD) — 8-week manualized group-based behavioral intervention including compensatory cognitive training for difficulties with learning, memory, processing speed, executive functioning, verbal functioning, concentration, and attention.
  Other Names: Compensatory Cognitive Training
  Arms: Motivationally Enhanced Compensatory Cognitive Training for Major Depressive Disorder
Behavioral: Goal-focused Supportive Contact — 8-week group-based behavioral intervention primarily focused on setting and achieving short or long-term goals. Does not provide training in cognitive strategies, lifestyle strategies, or motivational enhancement.
  Arms: Goal-focused Supportive Contact

SUMMARY:
Individuals with depression often describe difficulties with memory, attention, concentration, and overall cognitive functioning, which can persist even after mood episodes get better, and can affect treatment and health outcomes.

The primary objective of this pilot clinical trial is to evaluate the feasibility and acceptability of a manualized, 8-week, Compensatory Cognitive Training (CCT) intervention for Veterans who received treatment for MDD in the past year and have persistent cognitive functioning deficits. The investigators will compare Motivationally Enhanced Compensatory Cognitive Training for Major Depressive Disorder (ME-CCT-MDD) to a robust comparator, Goal-focused Supportive Contact (GSC), to evaluate differences in outcome measures.

The investigators hypothesize that Motivationally Enhanced Compensatory Cognitive Training for Major Depressive Disorder (ME-CCT-MDD) will be feasible and acceptable to participants in a pilot trial of ME-CCT-MDD vs. Goal-focused supportive contact (GSC) for Veterans with recent MDD treatment and persistent cognitive symptoms.

This study will also evaluate the preliminary magnitude and direction of symptom change on measures of objective cognitive functioning, psychiatric symptomatology, psychosocial functioning, and quality of life.

The investigators hypothesize that CCT will improve objective cognitive functioning, psychiatric outcomes, psychosocial functioning, and quality of life in Veterans with recent MDD-related cognitive functioning deficits.

Participants who agree to participate in the study will:

1. Take part in an assessment of their cognition, symptoms, and functioning, which will take approximately 2 hours. The assessment will include an interview about their medical, psychiatric, and cognitive history. It will also include questionnaires about their symptoms and daily functioning as well as neuropsychological tests, which are paper-pencil tests that evaluate aspects of cognition such as memory, attention, and problem-solving skills.
2. Be randomly assigned (like the flip of a coin) to receive Goal-Focused Supportive Contact or Compensatory Cognitive Training. Both treatments will involve weekly groups with a mental health provider for approximately 2 hours per week for 8 weeks. Goal-Focused Treatment includes setting and achieving short-term and long-term goals for improving cognition and functioning. Compensatory Cognitive Training includes training in strategies to improve cognition and manage stress.
3. Complete a follow-up assessment of cognition, symptoms, and functioning 8 weeks after they begin treatment, as well as a brief interview about their experience in the group. These assessment sessions will take approximately 2 hours.

DETAILED DESCRIPTION:
Motivationally Enhanced Compensatory Cognitive Training for Major Depressive Disorder (ME-CCT-MDD) is a manualized group-based behavioral intervention (8 weeks, 2 hours per week) designed to improve cognitive functioning in Veterans with Major Depressive Disorder (MDD) and cognitive complaints. ME-CCT-MDD is an adaptation of CCT initially developed by clinicians and researchers at the VA Portland Healthcare System and the VA San Diego Healthcare System. CCT draws from the empirical and theoretical literature on compensatory strategy training for conditions characterized by cognitive complaints and impairments, including mild traumatic brain injury, psychosis, and mild cognitive impairment.

ME-CCT-MDD is a comprehensive treatment in that it addresses multiple types of symptoms and concerns that interfere with recovery from depressed mood episodes - cognitive impairments, neuropsychiatric symptoms, and lifestyle patterns that increase the risk of cognitive impairment, poor health, and MDD relapse. In addition to training in compensatory cognitive skills, ME-CCT-MDD includes mindfulness practices and motivational interviewing techniques to boost the adoption of lifestyle strategies (e.g., nutrition, exercise) that improve cognition and overall health. ME-CCT-MDD is designed to be easy to administer and as an adjunct to standard MDD treatment programs.

Given the high rate of MDD among Veterans, the prevalence of cognitive impairments among those with MDD, and the negative impact of cognitive impairments on vocational functioning, psychosocial functioning, quality of life, and treatment outcomes, an evidence-based cognitive training intervention that optimally addresses the complex needs of Veterans with MDD and cognitive impairments is of critical importance. This study will allow the investigators to assess the feasibility and acceptability of the ME-CCT-MDD intervention in preparation for a larger-scale pilot randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

1. Veterans 18 years of age or older
2. Self-reported concerns about cognitive functioning deficits or clinical concerns about cognitive functioning deficits documented in EHR
3. meets DSM-5 criteria for MDD and receiving treatment for this diagnosis at the Portland VA within the past year
4. moderate or greater depressive symptoms as assessed by a PHQ-9 score ≥ 10
5. current cognitive functioning deficits as determined by performance on at least two measures in one cognitive domain (i.e., memory, attention/processing speed, language, executive functioning) falling ≥1 SD below their age-appropriate norms in the absence of memory impairment.

Exclusion Criteria:

1. impaired capacity to understand study risks and benefits
2. history of TBI as defined by American College of Rehabilitation Medicine and VA/DoD criteria
3. meets DSM-5 criteria for a substance use disorder other than nicotine use disorder in the past 6 months
4. meets DSM-5 criteria for dementia, psychotic disorder, or "with psychotic features" specifier
5. active suicidal intent with significant clinical risk
6. auditory or visual impairments that would prevent ability to participate in cognitive rehabilitation group or assessments. Eligibility will be established by electronic medical record review conducted by study staff and will be confirmed by the Veteran during the initial phone call.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | From enrollment to the end of treatment at 8 weeks
  Number of participants included from eligible Veterans; Recruitment will be deemed feasible if investigators successfully screen 50% of Veterans referred to the study for eligibility and enroll 75% of screened Veterans who meet all study inclusion criteria.
Study Retention | From enrollment to the second assessment (within 2 weeks post-treatment)
  Retention will be deemed successful if the investigators achieve 80% completion for post-treatment assessments.
Rate of Intervention Completion | From enrollment to the end of treatment at 8 weeks
  Percentage of participants that complete the 8-week intervention.
Feasibility of Testing Procedures | From enrollment to the second assessment (within 2 weeks post-treatment)
  Percentage of participants where follow-up visit was completed.
Feasibility of data collection methods | From enrollment to the second assessment (within 2 weeks post-treatment)
  Percentage of participants with complete data sets.
Acceptability, by participant report | From enrollment to the second assessment (within 2 weeks post-treatment)
  Treatment will be deemed acceptable if ≥ 70% of Veterans score ≥ 12 on the Acceptability of Intervention Measure (AIM).

SECONDARY OUTCOMES:
Objective Cognitive Functioning, Pre-Post Change: WAIS-IV Digit Span Subtest (Overall) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests to assess pre-post differences in neuropsychological testing performance on the Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV): Digit Span Subtest (Overall).
  Per best neuropsychological testing practices, and standardized scoring procedures, participants' raw test scores are converted to a Scaled Score (SS) using age-adjusted normative samples. SS ranges from 1 to 19 (Mean=10, Standard Deviation=3) with higher scores indicating stronger relative performance.
Objective Cognitive Functioning, Pre-Post Change: WAIS-IV Digit Span Subtest (Digit Span Forward) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests to assess pre-post differences in neuropsychological testing performance on the Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV): Digit Span Subtest (Digit Span Forward).
  Per best neuropsychological testing practices, and standardized scoring procedures, participants' raw test scores are converted to a Scaled Score (SS) using age-adjusted normative samples. SS ranges from 1 to 19 (Mean=10, Standard Deviation=3) with higher scores indicating stronger relative performance.
Objective Cognitive Functioning, Pre-Post Change: WAIS-IV Digit Span Subtest (Digit Span Backward) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests to assess pre-post differences in neuropsychological testing performance on the Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV): Digit Span Subtest (Digit Span Backward).
  Per best neuropsychological testing practices, and standardized scoring procedures, participants' raw test scores are converted to a Scaled Score (SS) using age-adjusted normative samples. SS ranges from 1 to 19 (Mean=10, Standard Deviation=3) with higher scores indicating stronger relative performance.
Objective Cognitive Functioning, Pre-Post Change: WAIS-IV Digit Span Subtest (Digit Span Sequencing) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests to assess pre-post differences in neuropsychological testing performance on the Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV): Digit Span Subtest (Digit Span Sequencing).
  Per best neuropsychological testing practices, and standardized scoring procedures, participants' raw test scores are converted to a Scaled Score (SS) using age-adjusted normative samples. SS ranges from 1 to 19 (Mean=10, Standard Deviation=3) with higher scores indicating stronger relative performance.
Objective Cognitive Functioning, Pre-Post Change: WAIS-IV Coding | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests to assess pre-post differences in neuropsychological testing performance on the Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV): Coding.
  Per best neuropsychological testing practices, and standardized scoring procedures, participants' raw test scores are converted to a Scaled Score (SS) using age-adjusted normative samples. SS ranges from 1 to 19 (Mean=10, Standard Deviation=3) with higher scores indicating stronger relative performance.
Objective Cognitive Functioning, Pre-Post Change: WAIS-IV Symbol Search | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests to assess pre-post differences in neuropsychological testing performance on the Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV): Symbol Search.
  Per best neuropsychological testing practices, and standardized scoring procedures, participants' raw test scores are converted to a Scaled Score (SS) using age-adjusted normative samples. SS ranges from 1 to 19 (Mean=10, Standard Deviation=3) with higher scores indicating stronger relative performance.
Objective Cognitive Functioning, Pre-Post Change: CVLT-3 (Trials 1-5 Correct) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests to assess pre-post differences in neuropsychological testing performance on the California Verbal Learning Test - Third Edition (CVLT-3): Trials 1-5 Correct.
  Per best neuropsychological testing practices, and standardized scoring procedures, participants' raw test scores are converted to a Standard Score (StdS) using age-adjusted normative samples. StdS ranges from 40 to 160 (Mean=100, Standard Deviation=15) with higher scores indicating stronger relative performance.
Objective Cognitive Functioning, Pre-Post Change: CVLT-3 (Delayed Recall Correct) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests to assess pre-post differences in neuropsychological testing performance on the California Verbal Learning Test - Third Edition (CVLT-3): Delayed Recall Correct.
  Per best neuropsychological testing practices, and standardized scoring procedures, participants' raw test scores are converted to a Standard Score (StdS) using age-adjusted normative samples. StdS ranges from 40 to 160 (Mean=100, Standard Deviation=15) with higher scores indicating stronger relative performance.
Objective Cognitive Functioning, Pre-Post Change: CVLT-3 (Total Recall Correct) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests to assess pre-post differences in neuropsychological testing performance on the California Verbal Learning Test - Third Edition (CVLT-3): Total Recall Correct.
  Per best neuropsychological testing practices, and standardized scoring procedures, participants' raw test scores are converted to a Standard Score (StdS) using age-adjusted normative samples. StdS ranges from 40 to 160 (Mean=100, Standard Deviation=15) with higher scores indicating stronger relative performance.
Objective Cognitive Functioning, Pre-Post Change: CVLT-3 (Short Delay Free Recall) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests to assess pre-post differences in neuropsychological testing performance on the California Verbal Learning Test - Third Edition (CVLT-3): Short Delay Free Recall.
  Per best neuropsychological testing practices, and standardized scoring procedures, participants' raw test scores are converted to a Scaled Score (SS) using age-adjusted normative samples. SS ranges from 1 to 19 (Mean=10, Standard Deviation= 3) with higher scores indicating stronger relative performance.
Objective Cognitive Functioning, Pre-Post Change: CVLT-3 (Short Delay Cued Recall) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests to assess pre-post differences in neuropsychological testing performance on the California Verbal Learning Test - Third Edition (CVLT-3): Short Delay Cued Recall.
  Per best neuropsychological testing practices, and standardized scoring procedures, participants' raw test scores are converted to a Scaled Score (SS) using age-adjusted normative samples. SS ranges from 1 to 19 (Mean=10, Standard Deviation= 3) with higher scores indicating stronger relative performance.
Objective Cognitive Functioning, Pre-Post Change: CVLT-3 (Long Delay Free Recall) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests to assess pre-post differences in neuropsychological testing performance on the California Verbal Learning Test - Third Edition (CVLT-3): Long Delay Free Recall.
  Per best neuropsychological testing practices, and standardized scoring procedures, participants' raw test scores are converted to a Scaled Score (SS) using age-adjusted normative samples. StdS ranges from 1 to 19 (Mean=10, Standard Deviation= 3) with higher scores indicating stronger relative performance.
Objective Cognitive Functioning, Pre-Post Change: CVLT-3 (Long Delay Cued Recall) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests to assess pre-post differences in neuropsychological testing performance on the California Verbal Learning Test - Third Edition (CVLT-3): Long Delay Cued Recall.
  Per best neuropsychological testing practices, and standardized scoring procedures, participants' raw test scores are converted to a Scaled Score (SS) using age-adjusted normative samples. SS ranges from 1 to 19 (Mean=10, Standard Deviation= 3) with higher scores indicating stronger relative performance.
Objective Cognitive Functioning, Pre-Post Change: CVLT-3 (Recognition Discriminability) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests to assess pre-post differences in neuropsychological testing performance on the California Verbal Learning Test - Third Edition (CVLT-3): Recognition Discriminability.
  Per best neuropsychological testing practices, and standardized scoring procedures, participants' raw test scores are converted to a Scaled Score (SS) using age-adjusted normative samples. SS ranges from 1 to 19 (Mean=10, Standard Deviation= 3) with higher scores indicating stronger relative performance.
Objective Cognitive Functioning, Pre-Post Change: BVMT-R (Total Recall) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests to assess pre-post differences in neuropsychological testing performance on the Brief Visuospatial Memory Test - Revised (BVMTR): Total Recall.
  Per best neuropsychological testing practices, and standardized scoring procedures, participants' raw test scores are converted to a T-Score using age-adjusted normative samples. T-Scores range from 20 to 80 (Mean=50, Standard Deviation= 10) with higher scores indicating stronger relative performance.
Objective Cognitive Functioning, Pre-Post Change: BVMT-R (Delayed Recall) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests to assess pre-post differences in neuropsychological testing performance on the Brief Visuospatial Memory Test - Revised (BVMTR): Delayed Recall.
  Per best neuropsychological testing practices, and standardized scoring procedures, participants' raw test scores are converted to a T-Score using age-adjusted normative samples. T-Scores range from 20 to 80 (Mean=50, Standard Deviation= 10) with higher scores indicating stronger relative performance.
Objective Cognitive Functioning, Pre-Post Change: D-KEFS Verbal Fluency Test (Letter Fluency Total Correct) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests to assess pre-post differences in neuropsychological testing performance on the Delis-Kaplan Executive Functioning System (D-KEFS): Verbal Fluency Test (Letter Fluency Total Correct).
  Per best neuropsychological testing practices, and standardized scoring procedures, participants' raw test scores are converted to a Scaled Score (SS) using age-adjusted normative samples. SS ranges from 1 to 19 (Mean=10, Standard Deviation= 3) with higher scores indicating stronger relative performance.
Objective Cognitive Functioning, Pre-Post Change: D-KEFS Verbal Fluency Test (Category Fluency Total Correct) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests to assess pre-post differences in neuropsychological testing performance on the Delis-Kaplan Executive Functioning System (D-KEFS): Verbal Fluency Test (Category Fluency Total Correct).
  Per best neuropsychological testing practices, and standardized scoring procedures, participants' raw test scores are converted to a Scaled Score (SS) using age-adjusted normative samples. SS ranges from 1 to 19 (Mean=10, Standard Deviation= 3) with higher scores indicating stronger relative performance.
Objective Cognitive Functioning, Pre-Post Change: D-KEFS Verbal Fluency Test (Category Switching Total Correct) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests to assess pre-post differences in neuropsychological testing performance on the Delis-Kaplan Executive Functioning System (D-KEFS): Verbal Fluency Test (Category Switching Total Correct).
  Per best neuropsychological testing practices, and standardized scoring procedures, participants' raw test scores are converted to a Scaled Score (SS) using age-adjusted normative samples. SS ranges from 1 to 19 (Mean=10, Standard Deviation= 3) with higher scores indicating stronger relative performance.
Objective Cognitive Functioning, Pre-Post Change: D-KEFS Verbal Fluency Test (Category Switching Total Switching Accuracy) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests to assess pre-post differences in neuropsychological testing performance on the Delis-Kaplan Executive Functioning System (D-KEFS): Verbal Fluency Test (Category Switching Total Switching Accuracy).
  Per best neuropsychological testing practices, and standardized scoring procedures, participants' raw test scores are converted to a Scaled Score (SS) using age-adjusted normative samples. SS ranges from 1 to 19 (Mean=10, Standard Deviation= 3) with higher scores indicating stronger relative performance.
Objective Cognitive Functioning, Pre-Post Change: D-KEFS Trail Making Test (Visual Scanning) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests to assess pre-post differences in neuropsychological testing performance on the Delis-Kaplan Executive Functioning System (D-KEFS): Trail Making Test (Visual Scanning).
  Per best neuropsychological testing practices, and standardized scoring procedures, participants' raw test scores are converted to a Scaled Score (SS) using age-adjusted normative samples. SS ranges from 1 to 19 (Mean=10, Standard Deviation= 3) with higher scores indicating stronger relative performance.
Objective Cognitive Functioning, Pre-Post Change: D-KEFS Trail Making Test (Number Sequencing) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests to assess pre-post differences in neuropsychological testing performance on the Delis-Kaplan Executive Functioning System (D-KEFS): Trail Making Test (Number Sequencing).
  Per best neuropsychological testing practices, and standardized scoring procedures, participants' raw test scores are converted to a Scaled Score (SS) using age-adjusted normative samples. SS ranges from 1 to 19 (Mean=10, Standard Deviation= 3) with higher scores indicating stronger relative performance.
Objective Cognitive Functioning, Pre-Post Change: D-KEFS Trail Making Test (Letter Sequencing) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests to assess pre-post differences in neuropsychological testing performance on the Delis-Kaplan Executive Functioning System (D-KEFS): Trail Making Test (Letter Sequencing).
  Per best neuropsychological testing practices, and standardized scoring procedures, participants' raw test scores are converted to a Scaled Score (SS) using age-adjusted normative samples. SS ranges from 1 to 19 (Mean=10, Standard Deviation= 3) with higher scores indicating stronger relative performance.
Objective Cognitive Functioning, Pre-Post Change: D-KEFS Trail Making Test (Number-Letter Switching) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests to assess pre-post differences in neuropsychological testing performance on the Delis-Kaplan Executive Functioning System (D-KEFS): Trail Making Test (Number-Letter Switching).
  Per best neuropsychological testing practices, and standardized scoring procedures, participants' raw test scores are converted to a Scaled Score (SS) using age-adjusted normative samples. SS ranges from 1 to 19 (Mean=10, Standard Deviation= 3) with higher scores indicating stronger relative performance.
Objective Cognitive Functioning, Pre-Post Change: D-KEFS Trail Making Test (Motor Speed) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests to assess pre-post differences in neuropsychological testing performance on the Delis-Kaplan Executive Functioning System (D-KEFS): Trail Making Test (Motor Speed).
  Per best neuropsychological testing practices, and standardized scoring procedures, participants' raw test scores are converted to a Scaled Score (SS) using age-adjusted normative samples. SS ranges from 1 to 19 (Mean=10, Standard Deviation= 3) with higher scores indicating stronger relative performance.
Self-Report Measures, Pre-Post Symptom Change | From enrollment to the second assessment (within 2 weeks post-treatment)
  Self-Reported Psychiatric and Cognitive Symptomatology, Psychosocial Functioning, and Quality of Life; Pre-Post Symptom Change Magnitude and direction of symptom change will be assessed by examining pre-post differences on self-report measures.
  Questionnaire Battery Includes: Patient Health Questionnaire (PHQ-9), WHO Disability Assessment Schedule (WHODAS 2.0), Prospective-Retrospective Memory Questionnaire (PRMQ), Neuro-QOL: Cognition & Ability to Participate in Social Roles and Activities, Portland Cognitive Strategies Scale 2.0 (PCSS).
Self-Report Measures, Pre-Post Symptom Change: PHQ-9 | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests for evaluating pre-post differences in self-reported symptomatology on the Patient Health Questionnaire-9 (PHQ-9).
  Scores range from 0 to 27, with higher scores indicating greater symptom severity.
Self-Report Measures, Pre-Post Symptom Change: WHODAS 2.0 (General Disability Score) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests for evaluating pre-post differences in self-reported symptomatology on the WHO Disability Assessment Schedule 2.0 (WHODAS 2.0): General Disability Score.
  Scores range from 36 to 180, with higher scores indicating greater symptom severity.
Self-Report Measures, Pre-Post Symptom Change: Prospective-Retrospective Memory Questionnaire (PRMQ) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests for evaluating pre-post differences in self-reported symptomatology on the Prospective-Retrospective Memory Questionnaire (PRMQ).
  Scores range from 16 to 80, with higher scores indicating greater symptom severity.
Self-Report Measures, Pre-Post Symptom Change: Neuro-QoL (Cognition Subscale) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests for evaluating pre-post differences in self-reported symptomatology on the Quality of Life in Neurological Disorder (Neuro-QOL): Cognition Subscale
  Scores range from 28 to 140, with higher scores indicating greater functional ability.
Self-Report Measures, Pre-Post Symptom Change: Neuro-QoL (Ability to Participate in Social Roles and Activities Subscale) | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests for evaluating pre-post differences in self-reported symptomatology on the Quality of Life in Neurological Disorder (Neuro-QOL): Ability to Participate in Social Roles and Activities.
  Scores range from 8 to 40, with higher scores indicating greater functional ability.
Self-Report Measures, Pre-Post Symptom Change: PCSS | From enrollment to the second assessment (within 2 weeks post-treatment)
  Magnitude and direction of symptom change will be assessed using paired sample t-tests for evaluating pre-post differences in self-reported symptomatology on the Portland Cognitive Strategies Scale 2.0 (PCSS).
  Scores range from 0 to 60, with higher scores indicating greater cognitive strategy usage.

CONTACTS AND LOCATIONS:
Overall Officials: Maya O'Neil, PhD, Principal Investigator — Portland VA Medical Center; Joren Adams, Principal Investigator — Portland VA Medical Center
Locations (1):
- Portland VA Medical Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No